CLINICAL TRIAL: NCT05975060
Title: A Phase 2/3 Open-Label Study to Evaluate the Safety and Immunogenicity of an XBB.1.5 (Omicron Subvariant) SARS CoV-2 rS Vaccine Booster Dose in Previously mRNA COVID 19 Vaccinated and Baseline SARS CoV 2 Seropositive COVID-19 Vaccine Naïve Participants
Brief Title: A Study to Evaluate the Safety and Immunogenicity of an (Omicron Subvariant) COVID-19 Vaccine Booster Dose in Previously Vaccinated Participants and Unvaccinated Participants.
Acronym: COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2019nCoV-313
Record Dates: First submitted 2023-07-28; First posted 2023-08-03 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: COVID-19, XBB.1.5
MeSH Terms: conditions — COVID-19 | interventions — Immunization, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group-A XBB.1.5 Vaccine (Booster) (Experimental): The Monovalent [5 μg/50 μg] NVX-CoV2601 XBB.1.5 Vaccine (Booster)
  Interventions: Biological: XBB.1.5 Vaccine (Booster)
- Group-B The monovalent XBB.1.5 Vaccine (Single Dose). (Active Comparator): Group-B The monovalent [5 μg/50 μg] NVX-CoV2601 XBB.1.5 Vaccine (Single Dose).
  Interventions: Biological: XBB.1.5 Vaccine (single dose)

INTERVENTIONS:
Biological: XBB.1.5 Vaccine (Booster) — Omicron sub variant XBB.1.5 SARS-CoV-2 rS /Matrix-M Adjuvant the monovalent [5 μg/50 μg] NVX-CoV2601) XBB.1.5 Vaccine (Booster)
  Other Names: Omicron sub variant XBB.1.5 vaccine( booster) SARS-CoV-2 rS /Matrix-M Adjuvant
  Arms: Group-A XBB.1.5 Vaccine (Booster)
Biological: XBB.1.5 Vaccine (single dose) — Omicron sub variant XBB.1.5 SARS-CoV-2 rS /Matrix-M Adjuvant the monovalent [5 μg/50 μg] NVX-CoV2601) XBB.1.5 Vaccine ( single dose)
  Other Names: Omicron sub variant XBB.1.5 vaccine(single dose) SARS-CoV-2 rS /Matrix-M Adjuvant
  Arms: Group-B The monovalent XBB.1.5 Vaccine (Single Dose).

SUMMARY:
This is a Phase 2/3 open-label study to evaluate the safety and immunogenicity of a booster dose of the XBB.1.5 severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant (r) spike (S) protein nanoparticle vaccine (SARS-CoV-2 rS) adjuvanted with Matrix-M™ in previously mRNA COVID-19 vaccinated adult participants ≥18 years of age and baseline SARS CoV-2 seropositive COVID-19 vaccine naïve participants ≥18 years of age.

DETAILED DESCRIPTION:
Novavax, Inc. developed a recombinant prototype COVID-19 vaccine constructed from the full-length ancestral (Wuhan) SARS CoV-2 S glycoprotein (GP) adjuvanted with the saponin-based Matrix-M adjuvant (NVX-CoV2373). Subsequently, the SARS CoV 2 Omicron variant and subvariants emerged with enhanced transmissibility and the most significant number of mutations in any strain to date. Current evidence demonstrates that variant strain mutations such as those in the Omicron XBB.1.5 sublineage confer the ability to evade both natural and vaccine-induced neutralizing antibodies.

Part 1 of the study aims to investigate the safety and immunogenicity of the Novavax XBB.1.5 SARS-CoV-2 rS vaccine (NVX-CoV2601) adjuvanted with Matrix-M in previously COVID-19 mRNA vaccinated participants to determine if it induces superior antibody responses compared to a historical control of the prototype vaccine (original Wuhan strain), NVX-CoV2373.

Part 2 of the study aims to investigate the safety and immunogenicity of 1 dose of NVX CoV2601 in baseline SARS-CoV-2 seropositive COVID-19 vaccine naïve participants to determine if it induces non-inferior antibody responses compared to 1 booster dose of NVX-CoV2601 in previously COVID-19 mRNA vaccinated individuals participating in Part 1.

Part 1:

Approximately 330 previously mRNA COVID-19 vaccinated participants will receive a booster dose of XBB.1.5 Omicron subvariant vaccine (NVX-CoV2601) on Day 0. Immunogenicity and 28-day safety data will be used for an interim analysis, while participants remain on the study for immunogenicity and safety data collection up to Day 180 post-vaccination.

Part 2:

After completion of Part 1, approximately 330 unvaccinated participants with a clinical history of COVID-19-like disease during the previous year will receive a booster dose of NVX-CoV2601 on Day 0. Immunogenicity and 28-day safety data will be used for an interim analysis, while participants remain on the study for immunogenicity and safety data collection up to Day 180 post vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age at time of study vaccination.
2. Part 1: Previously vaccinated with ≥ 3 doses of the Moderna and/or Pfizer /BioNTech prototype monovalent and/or BA.4/5 containing bivalent COVID-19 vaccines with the last dose administered ≥ 90 days prior to study vaccination.

   Part 2: Clinical history of COVID-19-like disease during the previous year.
3. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
4. Female participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea ≥ 12 consecutive months]) must agree to be heterosexually in-active from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from ≥ 28 days prior to enrollment and through the end of the study.

   1. Condoms (male or female) with spermicide (if acceptable in country)
   2. Diaphragm with spermicide
   3. Cervical cap with spermicide
   4. Intrauterine device
   5. Oral or patch contraceptives
   6. Norplant®, Depo-Provera®, or other in country regulatory approved contraceptive method that is designed to protect against pregnancy.
   7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle NOTE: Periodic abstinence (eg, calendar, ovulation, sympto-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
5. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to study vaccination.
6. Agrees to not participate in any research involving receipt of investigational products (drug/biologic/device) including other SARS-CoV-2 prevention or treatment trials for the duration of the study.

NOTE: For participants who become hospitalized with COVID-19, participation in investigational treatment studies is permitted.

Exclusion Criteria:

1. Received COVID-19 vaccines other than Moderna and/or Pfizer-BioNTech in the past, inclusive of clinical trial COVID-19 vaccines.
2. Participation in research involving receipt of investigational products (drug/biologic/device) within 90 days prior to study vaccination (Day 0).
3. Received influenza vaccination within 14 days prior to study vaccination, or any other vaccine within 30 days prior to study vaccination.
4. Any known allergies to products contained in the investigational product.
5. Any history of anaphylaxis to any prior vaccine.
6. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy.

   NOTE: Stable endocrine disorders (eg, thyroiditis, pancreatitis), including stable diabetes mellitus with no history of diabetic ketoacidosis are NOT excluded.
7. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorti-coids, or other immune-modifying drugs within 90 days prior to study vaccination (Day 0).

   NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical or intranasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted. Use of inhaled glucocorticoids is prohibited.
8. Received any prohibited medication (see Section 7.4.1), immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to study vaccination (Day 0).
9. Active cancer (malignancy) on chemotherapy within 3 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo malign and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
10. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.
11. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to study vaccination that, in the opinion of the investigator, might interfere with protocol compliance.
12. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (includ-ing neurologic or psychiatric conditions likely to impair the quality of safety reporting).
13. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization [CRO], and study site personnel involved in the conduct or planning of the study).
14. Known history of myocarditis or pericarditis.
15. Respiratory symptoms in the past 3 days (ie, cough, sore throat, difficulty breathing).
16. Temperature of > 38°C within 24 hours of planned study vaccination (site measured or participant meas-ured).
17. Blood pressure of ≥ 160/100 mmHg.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 660 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Part 1: Pseudovirus neutralization (inhibitory dilution at a concentration of 50%; ID 50 ) to the NVX-CoV2601 vaccine | Day 28
  Pseudovirus neutralization (inhibitory dilution at a concentration of 50%; ID 50 ) to the NVX-CoV2601 vaccine assessed at Day 28 following study vaccination.
Part 1: Seroresponse Rates (SRRs) in ID 50 titers to the NVXCoV2601 vaccine | Day 28
  SRRs (proportion of seroconverted participants) in ID 50 titers to the NVXCoV2601 vaccine assessed at Day 28 following the study vaccination.
Part 2: SRRs in ID 50 titers to the XBB.1.5 Omicron subvariant | Day 28
  SRRs (proportion of seroconverted participants) in ID 50 titers to the XBB.1.5 Omicron subvariant assessed at Day 28 following study vaccination.
Part 2: ID 50 (Geometric Mean Titers) GMTs to the XBB.1.5 Omicron subvariant | Day 28
  ID 50 GMTs to the XBB.1.5 Omicron subvariant assessed at Day 28 following study vaccination.

SECONDARY OUTCOMES:
Part 1: Pseudovirus neutralization (inhibitory dilution at a concentration of 50%; ID50) to the NVX-CoV2601 vaccine | Day 28
  Pseudovirus neutralization (inhibitory dilution at a concentration of 50%; ID50) to the NVX-CoV2601 vaccine assessed at baseline and 28 days following study vaccination.
Part 1: ID 50 GMTs to the XBB.1.5 Omicron subvariant | Day 0 to Day 180
  ID 50 GMTs to the XBB.1.5 Omicron subvariant at relevant time points
Part 1: ID 50 geometric mean fold rise (GMFR) to the XBB.1.5 Omicron subvariant at relevant time points (Days 28 and 180) from baseline (Day 0). | Day 0 to Day 180
  ID 50 GMFR to the XBB.1.5 Omicron subvariant at relevant time points (Days 28 and 180) from baseline (Day 0).
Part 1: SRRs in ID 50 titer concentrations to the XBB.1.5 Omicron subvariant at relevant time points. | Day 28 to Day 180
  SRRs in ID 50 titer concentrations to the XBB.1.5 Omicron subvariant at relevant time points.
Part 1: Anti-S immunoglobulin G (IgG) geometric mean concentrations (GMCs, EU/mL) to the NVX-CoV2601 vaccine at relevant time points | Day 0 to Day 180
  Anti-S IgG geometric mean concentrations (GMCs, EU/mL) to the NVX-CoV2601 vaccine at relevant time points (Days 0, 28, and 180).
Part 1: Incidence and severity of solicited local and systemic adverse events (AEs) | Day 0 to Day 7
  Incidence, duration, and severity of solicited local and systemic adverse events (AEs) for 7 days following vaccination.
Part 1: Incidence and severity of unsolicited AEs | Day 28
  Incidence, severity, and relationship of unsolicited AEs through 28 days after vaccination.
Part 1: Incidence and severity of MAAEs attributed to study vaccine, adverse events of special interest (AESIs), and serious adverse events (SAEs) | Day 0 to Day 180
  Incidence and severity of Medically attended adverse event (MAAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) through day 180 or EOS.
Part 2: Pseudovirus neutralization (ID 50 ) to the XBB.1.5 Omicron subvariant | Day 0 to Day 28
  Pseudovirus neutralization (ID 50 ) to the XBB.1.5 Omicron subvariant assessed at baseline and at Day 28 following study vaccination.
Part 2: Incidence and severity of solicited local and systemic adverse events (AEs) | Day 0 to Day 7
  Incidence, duration, and severity of solicited local and systemic adverse events (AEs) for 7 days following vaccination.
Part 2: Incidence, and severity of unsolicited AEs | Day 28
  Incidence, severity, and relationship of unsolicited AEs through 28 days after vaccination.
Part 2: Incidence and severity of MAAEs, AESIs, and SAEs | Day 0 to Day 180
  Incidence and severity of MAAEs attributed to study vaccine, adverse events of special interest (AESIs) (predefined list including PIMMCs, myocarditis and/or pericarditis, and complications specific to COVID-19), and serious adverse events (SAEs) through day 180 or EOS.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (30):
- United States (30):
  - AMR, Mobile, Alabama
  - Benchmark Research, Sacramento, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - AMR LLC-Miami, Coral Gables, Florida
  - AMR, Fort Myers, Florida
  - Health Awareness,LLC, Jupiter, Florida
  - Tekton Research, Lawrenceville, Georgia
  - Alliance for Multispecialty RSCH, Newton, Kansas
  - Tekton Research, Wichita, Kansas
  - AMR New Orleans, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - AMR, Kansas City, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Velocity Clinical Research, Norfolk, Nebraska
  - AMR, Las Vegas, Nevada
  - AXCES Research, Albuquerque, New Mexico
  - Rochester Clinical Research, Rochester, New York
  - Tekton Research, Yukon, Oklahoma
  - DM Clinical Research, Philadelphia, Pennsylvania
  - AMR, Knoxville, Tennessee
  - Benchmark Research, Austin, Texas
  - Tekton Research, Austin, Texas
  - Tekton Research, Beaumont, Texas
  - Pan American clinical Research,LLC, Brownsville, Texas
  - Benchmark Research, Fort Worth, Texas
  - Research For Your Health, Plano, Texas
  - Tekton Research, San Antonio, Texas
  - AMR Layton Research Centre, Layton, Utah
  - Health Research of Hampton Roads, Newport News, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Alves K, Kouassi A, Plested JS, Kalkeri R, Smith K, Kaba M, Nelson J, Zhu M, Cloney-Clark S, Cai Z, Mallory RM, Noriega F; 2019nCoV-313 Study Investigators. Immunogenicity and safety of a monovalent Omicron XBB.1.5 SARS-CoV-2 recombinant spike protein vaccine in previously unvaccinated, SARS-CoV-2 seropositive participants: Primary day-28 analysis of a phase 2/3 open-label study. Vaccine. 2025 May 10;55:127046. doi: 10.1016/j.vaccine.2025.127046. Epub 2025 Apr 2. PMID 40184816
- [Derived] Alves K, Kotloff K, McClelland RS, Kouassi A, Plested JS, Kalkeri R, Zhu M, Cloney-Clark S, Cai Z, Smith K, Kaba M, Nelson J, Hammershaimb EA, Mallory RM, Noriega F; 2019nCoV-313 Study Investigators. Immunogenicity and safety of a monovalent omicron XBB.1.5 SARS-CoV-2 recombinant spike protein vaccine as a heterologous booster dose in US adults: interim analysis of a single-arm phase 2/3 study. Lancet Infect Dis. 2025 May;25(5):585-594. doi: 10.1016/S1473-3099(24)00670-4. Epub 2025 Jan 14. PMID 39824198